CLINICAL TRIAL: NCT07052968
Title: Invasive and Non-invasive Haemodynamic Assessment of Pulmonary Hypertension in Chronic Kidney Disease Patient
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Randa Ahmed Sarhan, Dr,, Assiut University
Other Study IDs: RHC in PH pts e ckd
Record Dates: First submitted 2025-05-17; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Hypertension; Chronic Kidney Disease
MeSH Terms: conditions — Hypertension, Pulmonary; Renal Insufficiency, Chronic | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Echocardiography — Echocardiography is the non invasvive interventional assessment and the RHC is the invasive international assessment of the hemodynamics in PH patients with ckd.

SUMMARY:
Patients with CKD who suspected to have pulmonary hypertension by echocardiography with high probability, RHC used to confirm the diagnosis, assessment of hemodynamic parameters, differentiate pre and post capillary types of pulmonary hypertension and asses severity of the disease.

DETAILED DESCRIPTION:
Pulmonary Hypertension (PH ) is a haemodynamic and pathophysiological condition characterized by an increase in mean pulmonary arterial pressure ≥ 20 mmHg at rest, measured by right heart catheterization [1]. It results from various etiologies and multifactorial mechanisms. PH is associated with increased morbidity and mortality in patients with chronic kidney disease (CKD) .

CKD is defined as abnormalities in kidney structure or function persisting for more than three months, with implications for health. The latest KDIGO guidelines classify CKD based on glomerular filtration rate and albuminuria categories [2]. CKD has systemic complications a cardiovascular and pulmonary vascular disorders.

The PH in CKD patients is multifactorial, involving volume overload, endothelial dysfunction, vascular calcification, and increased left sided pressures [3].

Echocardiography is the primary non-invasive tool for assessing PH . It estimates systolic pulmonary artery pressure and evaluates right ventricular structure and function . Although widely accessible, ECHO has limitations ;operator dependency and potential underestimation or overestimation of pressures [4]. ESC/ERS guidelines for pulmonary hypertension in assessing the probablity (6) as :

High probability: TRV >3.4 m/s or TRV 2.9-3.4 m/s with other echo PH signs Intermediate probability: TRV 2.9-3.4 m/s without other echo PH signs Low probability: TRV ≤2.8 m/s and no other PH signs. Right heart catheterization (RHC) remains the gold standard for definitive PH diagnosis. It provides direct hemodynamic measurements, distinguishing pre-capillary from post-capillary PH. RHC is crucial for guiding targeted therapy and risk stratification, ensuring accurate management in CKD patients with suspected PH (5).

ELIGIBILITY:
Inclusion Criteria:

- All adult (aged 18 years old and older) patients who were diagnosed CKD(The presence of kidney damage or an estimated glomerular filtration rate (eGFR) of less than 60 mL/min/1.73 m², persisting for 3 months or more) and suspected to have pulmonary hypertension by clinical feature or by echocardiography with high probability were included in this study.

Exclusion Criteria:

* • Patients under 18 years old

  * Patient with chronic chest disease.
  * Patient bleeding diathesis and high risk of bleeding.
  * Individuals having acute kidney injury.
  * Patient developing other PH aetiologies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All genders
Study Population: Admitted patients in Internal medicine department, Critical care unit and pulmonary hypertension unit chest department at Assuit University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of pulmonary hypertention in chronic kidney diseaes patients and identify its type and guide management. | One year
  Hemodynamic assessment by echo including (right atrial surface area, right ventricular diameters, tricuspid annular plane systolic excursion ,tricusped regureg Jet velocity, inferior vena cava diameter and inspiratory collapability, estimated pulmonary artery pressure and left ventricular structure and function) and Hemodynamic assessment by RHC to diagnose and identify tyoe of PH according theses parameters a mean pulmonary arterial pressure (mPAP) >20 mm Hg, pulmonary artery wedge pressure (PAWP) ≤15mmHg and a PVR > 2WU. Pre-capillary PH ,mPAP >20 mmHg,PAWP ≤15mmHg,PVR ≥3WU.Isolated post-capillary PH (IpcPH),mPAP >20 mmHg,PAWP >15mmHg,PVR <3WU. Combined pre- and post-capillary PH (CpcPH),mPAP >20 mmHg,PAWP >15mmHg,PVR ≥3WU.Descriptive statistics will be done in the form of frequencies, mean and SD then analytic statistics will be done as chi square, independent sample test, correlations and regression tests, paired t-test will be

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jankowich M, Hebel R, Jantz J, Abbasi S, Choudhary G. Multispecialty pulmonary hypertension clinic in the VA. Pulm Circ. 2017 Oct-Dec;7(4):758-767. doi: 10.1177/2045893217726063. Epub 2017 Aug 22. PMID 28770656
- [Background] Pugh ME, Hemnes AR, Trammell A, Newman JH, Robbins IM. Variability in hemodynamic evaluation of pulmonary hypertension at large referral centers. Pulm Circ. 2014 Dec;4(4):679-84. doi: 10.1086/678514. PMID 25610603